CLINICAL TRIAL: NCT04623086
Title: A Randomized Comparison of Transitioning From Insulin GLargine to Insulin Degludec usING a Bridging Dose of Glargine Versus Direct Conversion, in Patients With Type 1 Diabetes Mellitus - a Pilot Study
Brief Title: Comparison of Glargine to Degludec Insulin Transition With or Without a Bridging Glargine Dose
Acronym: GLIDING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Arthi Thirumalai, Assistant Professor, School of Medicine: Metabolism, Endocrinology and Nutrition, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00008108
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: Insulin glargine, insulin degludec
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Glargine and Insulin Degludec (Experimental): Insulin glargine, 100 units per mL injected subcutaneously daily Insulin Degludec, 100 units per mL injected subcutaneously daily
  Interventions: Drug: Insulin Degludec; Drug: Insulin Glargine
- Insulin Degludec and placebo (Placebo Comparator): Insulin Degludec, 100 units per mL injected subcutaneously daily Placebo, 9g/L sodium chloride (normal saline) injected subcutaneously daily
  Interventions: Drug: Insulin Degludec; Drug: Placebo

INTERVENTIONS:
Drug: Insulin Degludec — Insulin Degludec injection
  Other Names: Tresiba
Drug: Insulin Glargine — Insulin Glargine injection
  Other Names: Lantus
  Arms: Insulin Glargine and Insulin Degludec
Drug: Placebo — 9g/L sodium chloride (normal saline) subcutaneous injection manufactured to mimic insulin glargine injection
  Arms: Insulin Degludec and placebo

SUMMARY:
This study evaluates direct switching vs use of a bridging dose from insulin glargine to insulin degludec in type 1 DM patients. Half of the participants will receive a bridging insulin glargine dose along with the 1st dose of degludec, while other half will receive a placebo and 1st dose of degludec.

DETAILED DESCRIPTION:
Insulin degludec (IDeg), an ultra-long-acting basal insulin, is increasingly used to treat patients with type 1 diabetes (T1D). IDeg has a half-life of 25 hours and duration of action exceeding 42 hours in patients with T1D and as a result does not require as stringent a dosing schedule as other basal insulins. However, steady state concentration of IDeg is not reached until 2 to 3 doses are administered daily, and this may result in greater glycemic variability in the 24 to 72 hours following the initiation of therapy with IDeg.

Our hypothesis is that among patients who transition from insulin glargine to IDeg, those who use a bridging dose of insulin glargine will not have a significant change, on average, in time spent in target glycemic range during the transition period, whereas, those transitioning directly to IDeg will have a significant change in this parameter. We further hypothesize that those using the bridging dose of insulin glargine will have less hypoglycemia, less hyperglycemia and need fewer correction boluses than the direct-conversion patients during the transition period.

Though IDeg is being increasingly used in clinical practice, there are no guidelines on what is the best way to transition patients from other long-acting insulins, such as glargine, to IDeg. The package insert recommends 1:1 dose conversion from other basal insulins to IDeg, but this does not account for the time taken by IDeg to achieve steady state (typically 48-72 hours). There is no guidance on what to do in those 48-72 hours. Given the time taken for IDeg to achieve steady state, the period of transition from one insulin to another, can result in significant glycemic variation in the 24-72 hours after the first dose. We want to study how best to avoid or minimize this and the option of using a small dose of their original long-acting insulin has anecdotal evidence of success in our practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ALL inclusion criteria to be included in the study.

  1. Patient age is 18-75 years.
  2. Diagnosis of T1D of at least 1-year duration.
  3. Has the ability to provide informed consent before any trial-related activities.
  4. Treated with insulin glargine as their basal insulin in the 3 months preceding screening visit.
  5. Stable insulin regimen (defined as change of <20% in the total daily dose of insulin and no change to the basal insulin agent) over the 3 months preceding the screening visit.
  6. Patient willing to dose their basal insulin at bedtime.
  7. Hemoglobin A1c < 9% in the 3 months preceding screening visit.
  8. Able to self-administer their insulin doses.
  9. Able to do self-monitoring of blood glucose using a glucose meter and willing to do this at least 2 times daily for patients using a CGM that requires calibration prior to the study and 4 times daily for patients who were not using a CGM prior to the study.
  10. Agreeable to the use of a continuous glucose monitor (CGM) for the duration required in the study. If already using a CGM prior to the study, then agreeable to wearing the blinded study CGM concurrently during the study period.
  11. Will be reachable by phone and/or email to comply with study procedures.
  12. Will be able to comply with study procedures, per investigator's opinion.
  13. Patient agrees to not use correctional insulin unless BG ≥250 for the 48 hours before and after 1st dose of IDeg.

Exclusion Criteria:

* Patient must not have ANY of the exclusion criteria to be included in the study.

  1. Patients with eGFR <30 on at least 2 measurements within 1-year of the screening visit.
  2. History of myocardial infarction within 6 months preceding the screening visit.
  3. Patients taking non-insulin medications for the glycemic management of T1D (including metformin, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT-2 inhibitors, thiazolidinediones, alpha-glucosidase inhibitors, pramlintide)
  4. Known or suspected allergy to IDeg or one of its excipients.
  5. Pregnant, planning to become pregnant in the next 3 months or breastfeeding.
  6. Participation in a clinical trial with investigational drug within 1 month of the screening visit or at present.
  7. Skin condition that prevents the insertion of the CGM.
  8. Previously randomized and received drug in this study.
  9. Presence of decompensated or poorly controlled psychiatric conditions.
  10. Current known or suspected illicit substance use.
  11. Any anticipated surgery or procedure in the next 14 days.
  12. Patients using U-300 glargine as their basal insulin.
  13. Patients using insulin afrezza as their short-acting insulin.
  14. Use of glucocorticoid burst/pulse therapy within 14 days prior to screening visit (chronic stable glucocorticoid doses are acceptable).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthi Thirumalai, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medicine Diabetes Institute at South Lake Union, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 participants were screened, 37 were randomized, 37 completed the study.
Pre-assignment Details: 12 participants did not meet study inclusion/exclusion criteria and were screen failures. 47 participants started study procedures but only 37 were randomized.
Groups:
- Unassigned Group: Enrolled participants who discontinued the study prior to randomization to any treatment group
Period: Overall Study
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo | Unassigned Group
Started (I have now edited the numbers to reflect that only those who were assigned a treatment arm are included among "started". I have removed the ones who were either screen failures or withdrew consent prior to being assigned a treatment arm now.) | 19 | 18 | 10 (Enrolled participants who discontinued the study prior to randomization to any treatment group)
Completed | 19 | 18 | 0 (Enrolled participants who discontinued the study prior to randomization to any treatment group)
Not Completed | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: We included all participants who had completed the treatment period in the final analysis. This included wearing the study continuous glucose monitor from time of randomization to study completion and implementing the transition from baseline insulin regimen to degludec (3 doses at least) according to protocol. We did not include subjects who either were "Unassigned" or "Screen Failures" as we could not obtain all the baseline characteristics in these two groups of participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14) | 44 (16) | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 8 | 16 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 26 (21) | 17 (16) | 22 (19)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.7 (19.2) | 87.7 (23.6) | 80 (22.2)
Body mass index [Mean (Standard Deviation); unit: kilograms/meters squared] | 24.9 (6) | 27.1 (5) | 26 (5.4)
Hemoglobin A1c [Mean (Standard Deviation); unit: percent glycated hemoglobin] | 6.7 (0.6) | 6.9 (1) | 6.8 (0.8)
Total Daily Dose of Insulin [Mean (Standard Deviation); unit: Units/kilogram body weight/day] | 0.6 (0.2) | 0.8 (0.4) | 0.7 (0.3)
Creatinine [Mean (Standard Deviation); unit: milligrams/deciliter] | 0.82 (0.21) | 0.84 (0.1) | 0.83 (0.2)
Time in range (TIR) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent with blood glucose in 70-180 mg/dL range in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 65.4 (21.6) | 69.4 (17.2) | 67.4 (19.4)
Coefficient of Variation of Glucose [Mean (Standard Deviation); unit: percent of variation] | 31.1 (6.7) | 31.4 (8.3) | 31.2 (7.4)
Time above range-1 (TAR-1) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent with blood glucose in 180-250 mg/dL range in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 26.8 (17.2) | 19.4 (13.7) | 23.2 (15.9)
Time above range-2 (TAR-2) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent with blood glucose greater than 250 mg/dL range in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 5.5 (7.1) | 5.9 (8) | 5.7 (7.5)
Time below range-1 (TBR-1) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent with blood glucose in 54-70 mg/dL range in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 2.1 (2.1) | 4.1 (5.7) | 3 (4.3)
Time below range-2 (TBR-2) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent with blood glucose below 54 mg/dL range in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 0.3 (0.7) | 1.6 (5) | 0.9 (3.3)
Nocturnal time in range (N-TIR) [Mean (Standard Deviation); unit: percent of time measured] — Percent of time spent between midnight and 0600 hours on each night, with blood glucose in 70-180 mg/dL range, in the 48 hours prior to 1st dose of insulin degludec.
  percent of time measured | 60.3 (28.9) | 74.4 (25.5) | 67.2 (27.8)
Correction Boluses [Mean (Standard Deviation); unit: Number of boluses] — Number of correction boluses administered by patient in the 48 hours prior to 1st dose of insulin degludec.
  Number of boluses | 0.9 (1.2) | 1.5 (1.2) | 1.2 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Percent Time in Range
Description: Change in percent time spent in target glycemic range (TIR, glucose 70-180 mg/dL, both values included) in the 48 hours before and the 48 hours after the 1st dose of IDeg.
Time Frame: 48 hours prior to 48 hours after 1st dose of degludec insulin
Population: Change in percent time spent in target glycemic range (TIR, glucose 70-180 mg/dL, both values included) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 2 (14.7) | -6.1 (17.6)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; For our power calculations, we assumed the true change in TIR to be 0% for the bridging group and 15% for the direct-conversion group, and we assumed a common standard deviation of 15% (meaning the distributions of change in TIR are separated by 1 standard-deviation unit), and thereby obtained that 20 patients in each group would provide 87% power to observe a statistically significant (at the two-sided level of .05) difference in mean change of TIR; Test type: Other — Comparison of two groups; p = 0.14, t-test, 2 sided; Mean Difference (Net) = 8.1

2. Secondary Outcome: Coefficient of Variation (CV) of Percent-time-in-range
Description: Change in coefficient of variation of glucose (CV) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 48 hours prior to 48 hours after 1st dose of degludec insulin
Population: Change in coefficient of variation of glucose (CV) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Measure: Mean (Standard Deviation); unit: percent of variation
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percent of variation | 3 (6.9) | -1.1 (8.5)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p = 0.11, t-test, 2 sided; Mean Difference (Net) = 4.1

3. Secondary Outcome: Nocturnal Percent Time in Range of 70-180 mg/dL Nocturnal Time in Range (N-TIR)
Description: Change in nocturnal (defined as midnight to 0600 hours) time in range (glucose in 70-180 mg/dL range) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 4 days: Outcome Measure Time Frame 48 hours prior to 48 hours after 1st dose of degludec insulin
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 5.1 (34.6) | -7 (34.2)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p = 0.29, t-test, 2 sided; Mean Difference (Net) = 12.1

4. Secondary Outcome: Percent Time Above 180 mg/dL (TAR-1)
Description: Change in time above range (glucose in 181-250 mg/dL range, TAR-1) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 5.4 (15.4) | 6.5 (12.4)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p = 0.015, t-test, 2 sided; Mean Difference (Net) = -11.9

5. Secondary Outcome: Time Above Range-2 (TAR-2)
Description: Change in time above range (glucose above 250 mg/dL range, TAR-2) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 2.2 (6.8) | 1.9 (6.2)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other; p = 0.88, t-test, 2 sided; Mean Difference (Net) = 0.3

6. Secondary Outcome: Time Below Range-1 (TBR-1)
Description: Change in time below range (glucose 54-70 mg/dL range, TBR-1) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 48 hours prior to 48 hours after 1st dose of degludec insulin
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 1.1 (3.5) | -1.5 (3.4)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p = 0.031, t-test, 2 sided; Mean Difference (Net) = 2.6

7. Secondary Outcome: Time Below Range-2 (TBR-2)
Description: Change in time below range (glucose below 54 mg/dL range, TBR-2) in the 48 hours before and the 48 hours after the 1st dose of IDeg, as noted on study continuous glucose monitor (dexcom G6)
Time Frame: 48 hours prior to 48 hours after 1st dose of degludec insulin
Measure: Mean (Standard Deviation); unit: percentage of time in measured period
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 19 | 18
percentage of time in measured period | 0.3 (0.7) | -0.8 (4.2)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p = 0.27, t-test, 2 sided; Mean Difference (Net) = 1.1

8. Secondary Outcome: Correction Boluses
Description: Change in the number of daily correction boluses administered in the 48 hours before and 48 hours after the 1st dose of degludec insulin, as noted on insulin logs maintained by participants
Time Frame: 48 hours prior to 48 hours after 1st dose of degludec insulin
Measure: Mean (Standard Deviation); unit: boluses in 48 hours measured
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo
Number analyzed (Participants) | 17 | 16
boluses in 48 hours measured | 0 (1.0) | 0 (1.6)
Statistical Analysis 1: Comparison: Insulin Glargine and Insulin Degludec vs Insulin Degludec and Placebo; Test type: Other — Comparison of two groups; p > 0.99, t-test, 2 sided; Mean Difference (Net) = 0

ADVERSE EVENTS:
Time Frame: Screening visit through study completion (an average of 3 weeks).
Description: Non-Systematic
Groups:
- Insulin Glargine and Insulin Degludec: Insulin glargine, 100 units per mL injected subcutaneously daily Insulin Degludec, 100 units per mL injected subcutaneously daily
  Insulin Degludec: Insulin Degludec injection
  Insulin Glargine: Insulin Glargine injection
  Includes participants from randomization to treatment arm till study completion.
- Insulin Degludec and Placebo: Insulin Degludec, 100 units per mL injected subcutaneously daily Placebo, 9g/L sodium chloride (normal saline) injected subcutaneously daily
  Insulin Degludec: Insulin Degludec injection
  Placebo: 9g/L sodium chloride (normal saline) subcutaneous injection manufactured to mimic insulin glargine injection
  Includes participants from randomization to treatment arm till study completion.
- Entire Study Period: Includes all participants from screening visit till either study completion or study termination due to screen failure or withdrawal of consent
Arm/Group | Insulin Glargine and Insulin Degludec | Insulin Degludec and Placebo | Entire Study Period
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/59
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT04623086/Prot_SAP_002.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT04623086/ICF_003.pdf